CLINICAL TRIAL: NCT00966602
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Drug-Drug Interaction Study of VX-809 and VX-770 in Healthy Subjects
Brief Title: Drug-Drug Interaction Study of VX-809 and VX-770 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Medical Monitor, Vertex Pharmaceuticals Incorporated
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX08-809-005
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — lumacaftor; ivacaftor

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Period 1 (Experimental)
  Interventions: Drug: VX-809; Drug: Placebo
- Treatment Period 2 (Experimental)
  Interventions: Drug: VX-770; Drug: Placebo
- Treatment Period 3 (Experimental)
  Interventions: Drug: VX-809 & VX-770; Drug: Placebo

INTERVENTIONS:
Drug: VX-809 — VX-809 capsule, once daily for 14 days
  Arms: Treatment Period 1
Drug: VX-770 — VX-770 tablet, once every 12 hours for 14 days
  Arms: Treatment Period 2
Drug: VX-809 & VX-770 — VX-809 capsule, once daily, and VX-770 tablets, once every 12 hours, for 14 days
  Arms: Treatment Period 3
Drug: Placebo — Matching Placebo

SUMMARY:
The purpose of this study is to assess the pharmacokinetics and safety of co-administration of VX-770 and VX-809 in healthy adults.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an inherited disease resulting from defects to a gene known as the cystic fibrosis transmembrane conductance regulator (CFTR). CF affects approximately 70,000 children and adults worldwide (30,000 in the United States) and is the most common fatal genetic disease in persons of European descent. Despite progress in the treatment of CF with antibiotics and mucolytics, the predicted median age of survival for a person with CF is in the mid-30s. Though the disease affects multiple organs, most morbidity and mortality is caused by progressive loss of lung function.

This is a Phase 1, randomized, double-blind, placebo-controlled, multiple-dose study of orally administered VX-809 and VX-770 in healthy subjects. The study will evaluate safety and tolerability of co-administration of VX-809 and VX-770 in healthy volunteers.

Enrollment is planned for 24 subjects at 1 clinical site. Subjects will be randomized to receive study drug or placebo during three 14-day treatment periods separated by 14-day washout periods. In Treatment Period 1, subjects randomized to study drug will receive VX-809 every 24 hours. In Treatment Period 2, subjects randomized to study drug will receive VX-770 every 12 hours. In Treatment Period 3, subjects randomized to study drug will receive VX-809 every 24 hours and VX-770 every 12 hours. Subjects randomized to placebo will receive placebo during all treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject between 18 and 55 years of age, inclusive
* Body mass index (BMI) between 18.5 and 30.0 kg/m2, inclusive
* Subjects of child-bearing potential and who are sexually active must meet contraception requirements
* Female subject must have a negative serum pregnancy test at screening, Day -1, and throughout the study

Exclusion Criteria:

* History of any illness that, in the opinion of the investigator might confound the results of the study or pose an additional risk in administering study drug to the subject. This may include but is not limited to a significant history of cardiovascular, central nervous system, hepatobiliary or renal disease, or a history of mental illness
* Participated in a clinical study involving administration of either an investigational or a marketed drug within 60 days or 7 terminal half-lives (whichever is longer) before the Screening visit
* Subject who has received VX-770 or VX-809 in a previous clinical study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameters of VX-770 and its metabolites in plasma in the presence and absence of VX-809 | 70 days
PK parameters of VX-809 in plasma in the presence and absence of VX-770 | 70 days

SECONDARY OUTCOMES:
Safety as measured by adverse events, physical examination, and clinically significant changes in laboratory values (hematology, chemistry, coagulation, and urinalysis), electrocardiograms (ECGs), and vital signs. | 70 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (1):
- Zuidlaren, Netherlands